CLINICAL TRIAL: NCT06303388
Title: Effects of Bruegger's Exercises Versus Egoscue Exercise on Lower Cross Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/01721
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lower Cross Syndrome
Keywords: Pain; Hyperlordosis; Anterior pelvic tilt
MeSH Terms: conditions — Pain; Swayback

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egoscue Exercise (Experimental): • The Egoscue exercise comprise of 10 exercises which Included
  1. Static back alone and with breathing.
  2. Abdominal contraction while in the static back position.
  3. abductor press
  4. overhead extension
  5. elbow curls on a wall
  6. static wall
  7. upper spinal twist 8 pelvic tilts
  9.supine groin progressive 10.air bench exercises.
  Interventions: Other: Egoscue Exercise
- Bruegger's Exercise (Active Comparator): steps include in Breugger's Exercise
  1. Sit with your buttocks at the edge of a chair.
  2. Spread your legs apart slightly.
  3. Turn your toes out slightly.
  4. Rest your weight on your legs/feet & relax your abdominal muscles.
  5. Tilt your pelvis forward (i.e. arch your lower back) while lifting your chest up
  6. Rotate your arms outward while turning your palms up.
  7. Hold your head high in the air, with a slight arch in the neck. The patient is to slowly exhale by breathing out through their lips while actively externally rotating their arms and spreading their fingers. The patient is to perform this exercise once or twice every 20-30 minutes of prolonged sitting and held in this position for 30-60 seconds
  Interventions: Other: Bruegger,s Exercise

INTERVENTIONS:
Other: Bruegger,s Exercise — Bruegger's Exercise protocol along with conventional Physiotherapy.
  Arms: Bruegger's Exercise
Other: Egoscue Exercise — Egoscue Exercise along with conventional Physiotherapy.
  Arms: Egoscue Exercise

SUMMARY:
This study aims to find effects of Bruegger's Exercise versus Egoscue exercise on pain and hyperlordosis on patient with lower cross syndrome. This is interventional study which recruits 34 participants ,14 in each group.

DETAILED DESCRIPTION:
A randomized control trial will be conducted on patients with lower cross syndrome. A total number of 34 participants will be randomised into two groups with 17 participants in each group. Both groups will receive Hot Packs on the lumbar area for 10 minutes. Group A will receive Conventional Therapy and will follow protocol of Bruegger's Exercise. Group B will follow protocol of the Egoscue exercise. This study aims to decrease pain and hyperlordosis.

Each group will be assessed at baseline which will include pain through NPRS, hyperlordosis through flexicurve ruler and anterior pelvic tilt through pelvic inclinometer. Data from both groups will again be assessed after 4 weeks of intervention.

Protocol of Bruegger's Exercise: Pt. position: Upright sitting on a chair.

1. Sit with your buttocks at the edge of a chair.
2. Spread your legs apart slightly.
3. Turn your toes out slightly.
4. Rest your weight on your legs/feet & relax your abdominal muscles.
5. Tilt your pelvis forward (i.e. arch your lower back) while lifting your chest up
6. Rotate your arms outward while turning your palms up.
7. Hold your head high in the air, with a slight arch in the neck.

The patient is to perform this exercise once or twice every 20-30 minutes of prolonged sitting and held in this position for 30-60 seconds. To avoid non-compliance patient will be asked to perform five repetitions of particular exercise with five second hold during their clinical session.

Protocol of Egoscue Exercise The Egoscue group received a total of 10 exercises which includes

1. Static back alone and with breathing
2. Abdominal contraction while in the static back position
3. abductor press
4. Overhead extension
5. elbow curls on a wall
6. Static wall
7. Upper spinal twist
8. pelvic tilts
9. supine groin progressive
10. Air bench exercises

Week 1: 3 times with 10 s hold time Week 2: 5 times with 10 s hold time Week 3: 15 times with 10 s hold time Week 4: 20 times with 10 s hold time

ELIGIBILITY:
Inclusion Criteria: • Females and males aged between 16 to 65 years

* Participants had to present with low back pain
* Participants had to meet the criteria for lower crossed syndrome indicating tight hip flexors (Modified Thomas test) and erector spinae (visual assessment through toe touching) together with weak glutei (Prone Hip Extension Co-ordination/Strength Test) and abdominals (Trunk Flexion Co-ordination and Strength Test)and thoracic kyphosis.
* Angle of anterior pelvic tilt > 10 degrees

Exclusion Criteria: • Participants who would be undergoing other forms of treatment that may interfere with the study, for the duration of the study, including other manipulative and physical therapies specific to back pain.

* Presence of other conditions that may mimic low back pain, e.g. nerve entrapment.
* Participants taking any medication that may interfere with the results of this study including, pain medication, anti-inflammatory medication, and muscle relaxants.
* Surgery on the back, pelvis, or sacrum is indicated or has previously occurred
* LBP having localised or radiating pain.
* Practiced any kind of exercise or sports activity during the last 6 months.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Flexicurve Ruler | 12 day
  The flexicurve ruler (flexible) is commonly used to measure the degree of spinal curvature of the lumbar lordosis in the sagittal plane. The flexible ruler was placed according to the Youdas method, over spinous processes from T12 to S2 vertebrae. The ruler was then cautiously removed from the spine and traced onto a plain piece of white paper. A vertical line was drawn to connect the T12 and S2 landmarks (L line) and together with the maximum width of the lumbar curvature (H line
Pelvic Inclinometer | 12 day
  A pelvic inclinometer was used to measure the anterior/posterior inclination of the pelvis of the subjects. An inclinometer has a 23 Cm length base and two 15 Cm arms in each side that freely move 360 degrees in horizontal plane. The ends of the arms are placed on the bony landmarks.The subject was asked to stand with the feet shoulder width apart. Even pressure was applied to both the arms of the inclinometer at anterior superior iliac spine and posterior superior iliac spine, with a bubble in the center the reading was then measured in degrees.
NPRS | 12 Day
  Several pain scales are used clinically to evaluate the severity of musculoskeletal pain, one of which is the Numeric Pain Rating Scale (NPRS-11), which is an eleven-point scale in which the endpoints are the extremes of no pain at all (score of 0) and the worst pain the patient has ever experienced (score of 10).

SECONDARY OUTCOMES:
Modified Thomas Test | 12 day
  This test was performed with the patient supine and the thighs positioned over the edge of the examining table. The patient was told to grasp the thigh of the untested limb and pull it toward the chest to flatten the back and stabilise the pelvis, preventing an increase in lumbar lordosis. A standard stretch position for the iliopsoas muscle is demonstrated with the hip extended and the leg hanging freely with normal knee flexion. A positive test was indicated if the hip remained flexed against gravity on tested limb. Additionally, if there was also knee extension on the tested limb then further testing was needed to decide between a tight iliopsoas or rectus femoris muscle. This was done by passively extending the knee of the tested limb to neutralize the effect of the rectus femoris and find if there was still no change in hip flexion.
Visual Assessment through toe touching | 12 day
  The patient was seated on the examining table with the pelvis in a vertical position and the legs extended. The patient was asked to actively flex foreword in order to bring the forehead to the knees. The normal functioning of the erector spinae should display an even 'C' shaped curve and a distance of 10cm from the knees to the forehead. There should be also no knee flexion and involve no pelvic tilting. Any deviation from these norms indicates shortness of the erector spinae muscles.
Prone Hip Extension Co-ordination Test | 12 day
  The patient lay prone and raised the tested thigh into extension with the knee held in an extended position. The researcher then palpated the lumbar erector spinae and gluteus maximus muscles. A normal activation sequence was then observed and palpated which involved first the hamstring and gluteus maximus muscles, then the contralateral lumbar erector spinae muscles and lastly the ipsilateral lumbar erector spinae muscles. A positive test result occurred if the lumbar erector spinae contracted before the gluteus maximus muscles did.
Trunk Flexion Co-ordination and Strength Test | 12 day
  The patient lay supine with the arms either behind the neck or forward across the body and knees bent. The researcher then contacted the patient's heels or positioned a hand under the patient's lumbar spine. The patient was then asked to complete a posterior pelvic tilt and raise the trunk up until the scapulae cleared the table. This position was maintained for 2 seconds. The patient then held the pelvic tilt while lowering their back to the table. The patient was then instructed to perform 10 repetitions while holding the last repetition for 30 seconds. A positive test result occurred if the patient could not perform 10 repetitions without the lumbar spine or heels rising off the table.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ishtiaq, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waters T. The effect of Bruegger's exercise on chronic low back pain in association with lower crossed syndrome: University of Johannesburg (South Africa); 2014.
- [Background] Koes BW, van Tulder MW, Thomas S. Diagnosis and treatment of low back pain. BMJ. 2006 Jun 17;332(7555):1430-4. doi: 10.1136/bmj.332.7555.1430. No abstract available. PMID 16777886
- [Background] May S, Johnson R. Stabilisation exercises for low back pain: a systematic review. Physiotherapy. 2008;94(3):179-89
- [Background] Nourbakhsh MR, Arabloo AM, Salavati M. The relationship between pelvic cross syndrome and chronic low back pain. Journal of back and musculoskeletal rehabilitation. 2006;19(4):119-28.
- [Background] Kudchadkar GS, Gurudut P, Welling A. Comparative effect of mat pilates and egoscue exercises in asymptomatic individuals with lumbar hyperlordosis: A randomized controlled trial. Indian Journal of Physical Therapy and Research. 2019;1(2):79-88.
- [Background] Sequeira S, Gurudut P, Kage V. Exploring effects of Egoscue versus lumbar stabilisation exercises for lower crossed syndrome on postural stability and hyperlordotic posture correction. Comparative Exercise Physiology. 2023:1-12.
- [Background] Vehrs Z. The Effect of Egoscue Corrective Exercises on Chronic Knee and Hip Pain: Brigham Young University; 2014.
- [Background] Laxmi V R, G N, V S, G M, Gopinath Y, G T. Efficacy of Janda's approach versus bruegger's exercise in pelvic cross syndrome and its impact on quality of life. International Journal of Research in Pharmaceutical Sciences. 2020;11:1701-6.
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Kahl C, Cleland JA. Visual analogue scale, numeric pain rating scale and the McGill pain Questionnaire: an overview of psychometric properties. Physical therapy reviews. 2005;10(2):123-8.
- [Background] Macintyre NJ, Bennett L, Bonnyman AM, Stratford PW. Optimizing reliability of digital inclinometer and flexicurve ruler measures of spine curvatures in postmenopausal women with osteoporosis of the spine: an illustration of the use of generalizability theory. ISRN Rheumatol. 2011;2011:571698. doi: 10.5402/2011/571698. Epub 2011 Feb 7. PMID 22482067
- [Background] Khan N, Nouman M, Iqbal MA, Anwar K, Sajjad AG, Hussain SA. Comparing the Effect of Stretching and Muscle Energy Technique in the Management of Lower Cross Syndrome. Pakistan Journal of Medical & Health Sciences. 2022;16(07):31-